CLINICAL TRIAL: NCT06155279
Title: Phase II Study of Pembrolizumab in Combination With Cisplatin or Carboplatin and Pemetrexed as Induction Chemo+Immunotherapy in Resectable Epithelioid and Biphasic Pleural Mesothelioma (CHIMERA Study)
Brief Title: Induction Chemo+Immunotherapy in Resectable Epithelioid and Biphasic Pleural Mesothelioma (CHIMERA Study)
Acronym: CHIMERA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: MSD Italia S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOV-Me-01-2023-CHIMERA
Record Dates: First submitted 2023-11-22; First posted 2023-12-04 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Carboplatin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: The neoadjuvant systemic treatment will be based on three cycles of pembrolizumab 200 mg flat dose in combination with standard doses of cisplatin (75 mg/sm) or carboplatin (AUC 5) and pemetrexed (500 mg/sm) administered intra-venous every 3 weeks.
  The surgical intervention of pleurectomy/decortication will be planned to occur within 6 weeks after the completion of neoadjuvant treatment.
  The adjuvant systemic treatment will be based on 14 cycles of pembrolizumab 200 mg flat dose administered intra-venous every 3 weeks. Patients should be able to start pembrolizumab following surgery as soon as clinically feasible and within 10 weeks from surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm (Experimental): Single arm Carboplatin/Cisplatin - Pemetrexed - Pembrolizumab
  The neoadjuvant systemic treatment will be based on three cycles of pembrolizumab 200 mg flat dose in combination with standard doses of cisplatin (75 mg/sm) or carboplatin (AUC 5) and pemetrexed (500 mg/sm) administered intra-venous every 3 weeks.
  The surgical intervention of pleurectomy/decortication will be planned to occur within 6 weeks after the completion of neoadjuvant treatment.
  The adjuvant systemic treatment will be based on 14 cycles of pembrolizumab 200 mg flat dose administered intra-venous every 3 weeks. Patients should be able to start pembrolizumab following surgery as soon as clinically feasible and within 10 weeks from surgery.
  Interventions: Drug: Carboplatin/Cisplatin - Pemetrexed - Pembrolizumab

INTERVENTIONS:
Drug: Carboplatin/Cisplatin - Pemetrexed - Pembrolizumab — The neoadjuvant systemic treatment will be based on three cycles of pembrolizumab 200 mg flat dose in combination with standard doses of cisplatin (75 mg/sm) or carboplatin (AUC 5) and pemetrexed (500 mg/sm) administered intra-venous every 3 weeks.
  The surgical intervention of pleurectomy/decortication will be planned to occur within 6 weeks after the completion of neoadjuvant treatment.
  The adjuvant systemic treatment will be based on 14 cycles of pembrolizumab 200 mg flat dose administered intra-venous every 3 weeks. Patients should be able to start pembrolizumab following surgery as soon as clinically feasible and within 10 weeks from surgery.
  Other Names: Keytruda

SUMMARY:
This is a prospective, open-label, multi-site Phase II trial of pembrolizumab in combination with pemetrexed and cisplatin or carboplatin as neo-adjuvant therapy followed by surgery and adjuvant pembrolizumab in patients affected by resectable stage I-IIIa chemonaïve epithelioid/biphasic pleural mesothelioma.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-site Phase II trial of pembrolizumab in combination with pemetrexed and cisplatin or carboplatin as neo-adjuvant therapy followed by surgery and adjuvant pembrolizumab in patients affected by resectable stage I-IIIa chemonaïve epithelioid/biphasic pleural mesothelioma.

The neoadjuvant systemic treatment will be based on three cycles of pembrolizumab 200 mg flat dose in combination with standard doses of cisplatin (75 mg/sm) or carboplatin (AUC 5) and pemetrexed (500 mg/sm) administered intra-venous every 3 weeks.

The surgical intervention of pleurectomy/decortication will be planned to occur within 6 weeks after the completion of neoadjuvant treatment.

The adjuvant systemic treatment will be based on 14 cycles of pembrolizumab 200 mg flat dose administered intra-venous every 3 weeks. Patients should be able to start pembrolizumab following surgery as soon as clinically feasible and within 10 weeks from surgery.

All participating centers will enroll eligible patients and administer neoadjuvant and adjuvant systemic treatment.

Thoracic surgery will be centralized in two reference centres (AOUPD PADOVA AND HUMANITAS CANCER CENTER).

All eligible patients will undergo two multidisciplinary team discussions, before and after induction systemic treatment.

The primary objective of this trial is to determine the pathological complete response rate of pembrolizumab in combination with standard doses of cisplatin or carboplatin and pemetrexed administered intra-venous every 3 weeks for three cycles. Pathological response will be centrally assessed by a blinded pathologist.

Radiological and metabolic assessment through CT-scan and PET-CT will be performed at the baseline and at the end of neoadjuvant chemo-immunotherapy. Radiological CT-scan will be then performed every 9 weeks (+/- 1 week) during the adjuvant treatment. Further radiological follow-up after the end of study treatment (or for those patients with early treatment discontinuation without disease relapse) will be performed every 12 weeks until a two-year period from surgery, followed by every 18 weeks until the fifth year.

Radiological response will be centrally assessed by a blinded radiologist. Adverse events will be monitored throughout the trial and graded in severity according to the guidelines outlined in the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of surgical resectable stage I-IIIA treatment-naïve epithelioid/biphasic pleural mesothelioma will be enrolled in this study.
* Diagnosis of epithelioid/biphasic pleural mesothelioma must be histologically confirmed, preferably by video-assisted thoracoscopic surgery (VATS).
* At screening, complete surgical resection of the mesothelioma must be deemed achievable, as assessed by a multidisciplinary evaluation.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Measurable disease, defined as at least 1 lesion measured in two positions at three separate levels on transverse cuts of CT scan that is suitable for repeated assessment using modified Response Evaluation Criteria in Solid Tumours [m-RECIST 1.1] for pleural mesothelioma is preferred; however, inclusion of specific cases without measurable disease could be discussed with the medical monitor and during the multidisciplinary team discussion of the surgical centers.
* Histologically proved diagnosis of treatment-naive epithelioid/biphasic pleural mesothelioma.
* Surgical resectable disease [stage I - II - IIIA (T1-3 - N0/1-M0) according to ninth TNM edition].
* No previous surgical resection of mesothelioma.
* Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Has adequate PFT defined as an FEV1 >50% (of predicted normal volume) or ≥ 1.2 L/Sec and a DLCO >40% of predicted normal value. Participants for whom DLCO measurements are not available will be deemed to have adequate oxygen transfer if pulse oximetry (O2 saturation) ≥90% room air.
* Have adequate organ function as defined in the following table (Table 3). Specimens must be collected within 10 days prior to the start of study intervention.

Exclusion Criteria:

* Subject incapacitated to understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted
* Primitive peritoneal, pericardial and tunica vaginalis testis mesotheliomas.
* Cytological diagnosis of pleural mesothelioma not histologically confirmed.
* Prior treatment with systemic anti-cancer therapy for pleural mesothelioma, prior intraoperative intracavitary chemotherapy for pleural mesothelioma, prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Has uncontrolled, potentially reversible cardiac conditions, as Investigator's judgment (eg. Unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation > 500 millisecond) or participants with congenital long QT syndrome.
* Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-CNS disease is permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study intervention.
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
* Known additional malignancy that is progressing or has required active treatment within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or adequately treated carcinoma in-situ without evidence of disease are not excluded. Participants with low-risk early-stage prostate cancer (T1-T2a, Gleason score ≤6, and PSA <10 ng/mL) either treated with definitive intent or untreated in active surveillance with stable disease are not excluded.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid).
* History of Hepatitis B (defined as HbsAg reactive) or known active Hepatitis C virus (defined as detectable HCV RNA [qualitative]) infection.
* Has not adequately recovered from major surgery or has ongoing surgical complications.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.
* History of HIV infection. HIV testing is not required unless mandated by local health authority.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint - To evaluate the activity of neo-adjuvant treatment by the determination of pathological complete response rate (pCR) | Pathological complete response will be evaluated following neoadjuvant treatment and within 6 weeks after the last dose of study intervention.
  Pathological complete response defined as 0% residual viable tumor cells in the primary tumor and in sampled lymph nodes, following neoadjuvant treatment as assessed by central pathology assessment. Patients who are not evaluable per central pathology assessment (this includes patients with R2 margins) or who do not have a surgical specimen will be considered as non-pCR (eg, pathology assessments captured as "non-evaluable" or "missing," as appropriate). Patients who received less than 2 cycles out of the planned 3 cycles of neoadjuvant therapy due to unacceptable toxicity will not be considered in the pCR evaluation.

SECONDARY OUTCOMES:
Secondary endpoint - To further evaluate the activity of neo-adjuvant treatment in terms of major pathological response. | Major pathological response will be evaluated at the time of surgery that will be performed within 6 weeks after the last dose of study intervention.
  Major pathological response defined as ≤10% residual viable tumor cells in the primary tumor and sampled lymph nodes after neoadjuvant treatment at the time of resection as assessed per central pathology laboratory. Patients who are not evaluable per central pathology assessment (including patients with R2 margins) or who do not have a surgical specimen will be considered as having non-mPR (eg, response captured as "non-evaluable" or "missing," as appropriate).
Secondary endpoint - To further evaluate the activity of neo-adjuvant treatment in terms of overall response rate (ORR). | The ORR will be evaluated: at the time of the screening (within 4 weeks before the neoadjuvant treatment); within 6 weeks after neoadjuvant treatment; within 10 weeks after surgery; at every radiological assessment with CT-scan up to 24 months
  Overall response rate defined as the sum of partial and complete response according to modified RECIST 1.1 criteria for Malignant Pleural Mesothelioma.
Secondary endpoint - To evaluate the efficacy of neo-adjuvant treatment in terms of overall survival (OS). | From the start of treatment to death from any cause, up to 24 months.
  Overall survival defined as the time from the start of treatment to all-cause death.
Secondary endpoint - To evaluate the efficacy of neo-adjuvant treatment in terms of event free survival (EFS). | From the start of treatment to any progression of disease precluding surgery, progression or recurrence of disease after surgery, progression of disease in the absence of surgery, or death from any cause, up to 24 months.
  Event free survival defined as the time from the start of treatment to any progression of disease precluding surgery, progression or recurrence of disease after surgery, progression of disease in the absence of surgery, or death from any cause.
Secondary endpoint - To evaluate the feasibility of neo-adjuvant treatment in terms of resection rate and rate of patients who complete all cycles of neoadjuvant treatment and following surgery. | From the screening to the surgery which is performed within 6 weeks after the neoadjuvant treatment, up to 22 weeks.
  Feasibility in terms of: i) Resection rate: defined as the percentage of patients finally eligible for radical surgery, among those who receive at least one cycle of neoadjuvant treatment; ii) rate of patients who complete three cycles of neoadjuvant chemo-immunotherapy followed by radical surgery.
Secondary endpoint - To evaluate the safety profile of neoadjuvant treatment | Safety profile will be evaluated during the entire duration of the study, up to 24 months.
  Safety profile in terms of incidence and grade of adverse events; incidence of adverse events and serious adverse events; incidence of definitive interruptions of treatment because of any-cause adverse events and treatment-related adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Pasello, MD, Principal Investigator — Istituto Oncologico Veneto IOV IRCCS
Locations (8):
- Italy (8):
  - Humanitas Gavazzeni, Bergamo, Italia/Bergamo
  - IFO - Istituto Tumori Regina Elena, Roma, Roma, Italia/Roma
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Centro di Riferimento Oncologico (CRO) IRCCS, Aviano, Pordenone
  - Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliero-Universitaria S. Anna, Ferrara
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera-Universitaria di Parma, Parma

IPD SHARING:
Plan to Share IPD: No